CLINICAL TRIAL: NCT07066397
Title: A Phase 1 Study of Fast-In-Time Autologous Anti-CD19 Chimeric Antigen Receptor T Cells (FIT-CD19-CAR-T Cells) Infusion for Subjects With Relapsed/Refractory B-Cell Acute Lymphoblastic Leukemia
Brief Title: A Phase 1 Study of FIT-CD19-CAR-T Cells in R/R B-ALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TriArm Therapeutics (Taiwan) Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIT-CD19-CAR-T-003
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: CAR T-Cell Therapy; Acute lymphoblastic leukemia; CD19; non-viral; fast CAR
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ARM011 following lymphodepleting chemotherapy (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment with ARM011
  Interventions: Biological: ARM011; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: ARM011 — ARM011 is an autologous, CD19 targeted CAR T-cell product developed on fast-in-time (FIT) platform-a non-viral, 2-day rapid manufacturing process
Drug: Fludarabine — Administered prior to infusion of ARM011
Drug: Cyclophosphamide — Administered prior to infusion of ARM011

SUMMARY:
This is a Phase 1 study to evaluate FIT-CD19-CAR-T (ARM011) safety and tolerability, anti-tumor activity, cellular kinetics, immunogenicity, and exploratory biomarkers.

DETAILED DESCRIPTION:
This is an open-label, single arm, Phase 1 study to evaluate the safety and tolerability of FIT-CD19-CAR-T (ARM011) administered intravenously (IV) following a standard lymphodepleting (LD) chemotherapy regimen of cyclophosphamide and fludarabine in subjects with relapsed/refractory acute lymphoblastic leukemia (ALL). This dose finding study will use a 3+3 design.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subjects age ≥18 years
2. Diagnosis of ALL
3. Refractory to or relapsed after current standard treatment, and not suitable or unable to wait for other treatment options
4. Disease burden: Bone marrow with evidence of disease.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Adequate organ functions
7. Life expectancy ≥12 weeks

Key Exclusion Criteria:

1. Active central nervous system (CNS) involvement of ALL
2. Burkitt's lymphoma or chronic myeloid leukemia (CML) lymphoid blast crisis
3. Prior anti-CD19 therapy (other than blinatumomab)
4. Subjects who have experienced Grade 3 or higher cytokine release syndrome (CRS)/neurotoxicity following blinatumomab.
5. autoimmune disease resulting in end-organ injury or requiring systemic immunosuppression within the last 2 years.
6. History or presence of cardiac or CNS disorders as defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2041-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events [Safety and Tolerability] | Up to 24 months after ARM011 infusion
  Safety and Tolerability: Proportion of subjects experiencing adverse events and dose-limiting toxicities

SECONDARY OUTCOMES:
Evaluate cellular kinetics and persistence of ARM011 | Up to 24 months after ARM011 infusion
  Cellular kinetics related peak (Cmax) in peripheral blood
Evaluate cellular kinetics and persistence of ARM011 | Up to 24 months after ARM011 infusion
  Area under the concentration time curve (AUC) in peripheral blood
Evaluate preliminary anti-tumor activity of ARM011 | Up to 24 months after ARM011 infusion
  Preliminary anti-tumor activity: Proportion of subjects with an objective response (including complete response or complete remission with incomplete count recovery)
Evaluate host immunogenicity to ARM011 | Up to 24 months after ARM011 infusion
  Incidence of anti-CD19-directed CAR antibodies
Evaluate the feasibility of administration of ARM011 | 24 months
  The proportion of subjects for whom a CAR T-cell product meeting specifications could be prepared, which will be computed with a corresponding 95% confidence interval (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Hosein Kouros-Mehr, MD, PhD, Study Director — TriArm Inc.
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No